CLINICAL TRIAL: NCT01543360
Title: Comparison of Axillary Versus Subclavian Vein Strategies for Central Venous Catheterization Under Continuous Ultrasound Guidance: a Prospective, Randomized, Non-inferiority Study
Brief Title: Comparison of Axillary Versus Subclavian Vein Strategies for Central Venous Catheterization Under Continuous Ultrasound Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2011/JYL-GB-01; 2011-A01353-38 (Other: ANSM)
Record Dates: First submitted 2012-02-20; First posted 2012-03-05 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-03

CONDITIONS: Central Venous Catheterization
Keywords: axillary vein; sub clavian vein; comparison of strategies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axillary strategy (Active Comparator): The first two attempts at central venous catheterization will be performed via the distal approach (axillary vein). The third and fourth attempts at central venous catheterization will be performed by the medial approach (subclavian vein).
  Interventions: Procedure: Axillary strategy
- Subclavian strategy (Active Comparator): The first two attempts at central venous catheterization will be performed by the medial approach (subclavian vein). The third and fourth attempts at central venous catheterization will be performed by the distal approach (axillary vein).
  Interventions: Procedure: Subclavian strategy

INTERVENTIONS:
Procedure: Axillary strategy — The first two attempts at central venous catheterization will be performed via the distal approach (axillary vein). The third and fourth attempts at central venous catheterization will be performed by the medial approach (subclavian vein). The same puncture material/devices will be used in both arms of the study.
  Arms: Axillary strategy
Procedure: Subclavian strategy — The first two attempts at central venous catheterization will be performed by the medial approach (subclavian vein). The third and fourth attempts at central venous catheterization will be performed by the distal approach (axillary vein). The same puncture material/devices will be used in both arms of the study.
  Arms: Subclavian strategy

SUMMARY:
The main objective of this study is to compare the rate of successful establishment of a central venous catheter in the first two attempts of ultrasound-guided puncture between two techniques: (1) a subclavian technique versus (2) an axillary technique.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the following between the two techniques:

* the success rate of the establishment of a central venous catheter
* the success rate of establishment of a central venous catheter at the first attempt at venipuncture
* for non-failures (eg, a catheter is placed in the first four trys), time to cannulation
* the presence / absence of the following complications:
* arterial puncture (yes / no)
* pneumothorax (yes / no)
* hemothorax (yes / no)
* hematoma (yes / no)
* nerve injury (yes / no)
* aberrant course (yes / no)

The reasons catheter placement failures will also be described.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 24 hours of follow-up
* Patient requiring the establishment of a central venous catheter

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Patient has a body mass index < 15 or > 40
* Congenital or acquired anatomical deformity (radiation therapy, trauma, surgery) of the axillary and/or subclavian regions
* Bleeding disorder (platelets < 50,000, prothrombine < 50%, activated cephaline time > 2 times the control value)
* Severe hypoxemia defined by a ratio PaO2 / FIO2 < 100
* Infection of the puncture area
* Known thrombosis of the subclavian or axillary veins
* Scheduled length of hospitalization less than 24 hours
* Agitated or non-cooperative patient
* The patient has already been included in this study
* subclavian and axillary veins are not simultaneously echogenic on one or both sides (left and right).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05-23 (Actual); Study Completion 2013-05-23 (Actual)

PRIMARY OUTCOMES:
Central venous catheter established within first 2 puncture attempts | approximately 3 minutes
  yes/no

SECONDARY OUTCOMES:
Central venous catheter established upon first punction attempt | approximately 3 minutes
  yes/no
Establishment of a central venous catheter | approximately 3 minutes
  yes/no
The time necessary for the establishment of a central venous catheter | approximately 3 minutes
  For non-failures (ie establishment of a central venous catheter within 4 puncture attempts), the number of minutes necessary for the establishment of a central venous catheter
The time necessary for the establishment of a central venous catheter | approximately 3 minutes
  all cases, in minutes
presence/absence of complications | Day 1
  arterial puncture (yes / no), pneumothorax (yes / no), hemothorax (yes / no), hematoma (yes / no), nerve injury (yes / no), aberrant course (yes / no)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves Lefrant, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France

REFERENCES:
- [Result] Buzancais G, Roger C, Bastide S, Jeannes P, Lefrant JY, Muller L. Comparison of two ultrasound guided approaches for axillary vein catheterization: a randomized controlled non-inferiority trial. Br J Anaesth. 2016 Feb;116(2):215-22. doi: 10.1093/bja/aev458. PMID 26787790